CLINICAL TRIAL: NCT00960999
Title: A Randomized Phase II Study Comparing 2 Stereotactic Body Radiation Therapy (SBRT) Schedules for Medically Inoperable Patients With Stage I Peripheral Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy in Treating Patients With Stage I Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0915; CDR0000652101
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; squamous cell lung cancer; adenocarcinoma of the lung; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-fraction SBRT (34 Gy) (Experimental): Single-fraction stereotactic body radiation therapy (SBRT) of 34 Gy
  Interventions: Radiation: Single-fraction stereotactic body radiation therapy (SBRT)
- Multiple-fraction SBRT (48 Gy) (Experimental): Multiple-fraction stereotactic body radiation therapy (SBRT) given in four daily 12 Gy fractions for a total dose of 48 Gy
  Interventions: Radiation: Multiple-fraction stereotactic body radiation therapy (SBRT)

INTERVENTIONS:
Radiation: Single-fraction stereotactic body radiation therapy (SBRT) — 34 Gy in 1 fraction to the prescription line at the edge of the planning target volume (PTV). The maximum dose must exist within the PTV, and the prescription isodose surface must be ≥ 60% and < 90% of the maximum dose. 99% of the PTV must receive a minimum of 90% of the prescription dose. The maximum dose to any point ≥ 2 cm away from the PTV in any direction must be at least < 50% of the prescription dose. The percent of the lungs (excluding PTV) receiving 20 Gy or more must be < 10%.
  Arms: Single-fraction SBRT (34 Gy)
Radiation: Multiple-fraction stereotactic body radiation therapy (SBRT) — 48 Gy in four 12 Gy fractions to the prescription line at the edge of the planning target volume (PTV). Treatments are given on 4 consecutive calendar days, but at least 18 hours apart. The maximum dose must exist within the PTV, and the prescription isodose surface must be ≥ 60% and < 90% of the maximum dose. 99% of the PTV must receive a minimum of 90% of the prescription dose. The maximum dose to any point ≥ 2 cm away from the PTV in any direction must be at least < 50% of the prescription dose. The percent of the lungs (excluding PTV) receiving 20 Gy or more must be < 10%.
  Arms: Multiple-fraction SBRT (48 Gy)

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. It is not yet known which regimen of stereotactic body radiation therapy is more effective in treating patients with non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying the side effects of two radiation therapy regimens and to see how well they work in treating patients with stage I non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 1-year rate of ≥ grade 3 adverse events that are definitely, probably, or possibly related to treatment with single fraction vs multiple fraction stereotactic body radiotherapy in medically inoperable patients with stage I peripheral non-small cell lung cancer.

Secondary

* To estimate the 1-year primary tumor control rate in these patients.
* To estimate the 1-year overall survival and disease-free survival rate of these patients.
* To assess FDG-PET (fluorodeoxyglucose - positron emission tomography) standardized uptake value changes as a measure of treatment response and outcomes.
* To determine pulmonary function changes by treatment arm and response.
* To determine the association between biomarkers and primary tumor control and/or ≥ grade 2 radiation pneumonitis.

OUTLINE: This is a multicenter study. Patients are stratified according to Zubrod performance status (0 vs 1 vs 2) and T stage (T1 vs T2). Patients are randomized to 1 of 2 treatment arms.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation (by biopsy or cytology) of non-small cell lung cancer (NSCLC) prior to treatment; the following primary cancer types are eligible: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, large cell neuroendocrine, or non-small cell carcinoma not otherwise specified; Note: although bronchioloalveolar cell carcinoma is a subtype of NSCLC, patients with the pure type of this malignancy are excluded from this study because the spread of this cancer between adjacent airways is difficult to target on computed tomography (CT).
2. Stage T1, N0, M0 or T2 (≤ 5 cm), N0, M0, (AJCC Staging, 6th Ed.), based upon #3.
3. Minimum diagnostic workup:

   * History/physical examination, including weight and assessment of Zubrod performance status, within 4 weeks prior to registration;
   * Evaluation by an experienced thoracic cancer clinician (a thoracic surgeon, medical oncologist, radiation oncologist, or pulmonologist) within 8 weeks prior to registration;
   * CT scan with intravenous contrast (unless medically contraindicated) within 8 weeks prior to registration of the entirety of both lungs and the mediastinum, liver, and adrenal glands; the primary tumor dimension will be measured on the CT. Positron emission tomography (PET) evaluation of the liver and adrenal glands also is permitted. In addition, if the enrolling institution has a combined PET/CT scanner and both aspects are of diagnostic quality and read by a trained radiologist, the PET/CT will meet the staging requirements for both CT and PET.
   * Whole body or wide field FDG-PET within 8 weeks prior to registration with adequate visualization of the primary tumor and draining lymph node basins in the hilar and mediastinal regions and adrenal glands; in the event of lung consolidation, atelectasis, inflammation or other confounding features, PET-based imaging correlated with CT imaging will establish the maximal tumor dimensions. Standardized uptake value (SUV) must be measured on PET. To be included in this analysis, the patient's PET studies must be performed with a dedicated bismuth germanium oxide (BGO), lutetium oxyorthosilicate (LSO), or gadolinium oxyorthosilicate (GSO) PET or PET/CT scanner. PET scanners with sodium iodide (Nal) detectors are not acceptable. If the baseline PET study is performed at the treating institution (or its affiliated PET facility), it is recommended that the reassessment PET scans be performed at the same site.
   * Pulmonary function tests (PFTs): Routine spirometry, lung volumes, and diffusion capacity, within 8 weeks prior to registration; arterial blood gases are optional. Note: All patients enrolled in this study must have these pulmonary assessments whether or not the reason for their medical inoperability is pulmonary based, since the objective assessment of pulmonary factors is a component of the outcomes assessment for this study.
4. Patients with hilar or mediastinal lymph nodes ≤ 1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer.
5. The patient's resectable NSCLC must be considered medically inoperable by an experienced thoracic cancer clinician (a thoracic surgeon, medical oncologist, radiation oncologist, or pulmonologist) or a standard lobectomy and mediastinal lymph node dissection/sampling procedure. The patient may have underlying physiological medical problems that would prohibit a surgery due to a low probability of tolerating general anesthesia, the operation, the postoperative recovery period, or the removal of adjacent functioning lung. These types of patients with severe underlying health problems are deemed "medically inoperable." Standard justification for deeming a patient medically inoperable based on pulmonary function for surgical resection of NSCLC may include any of the following:

   * Baseline forced expiratory volume in one second (FEV1) < 40% predicted;
   * Postoperative FEV1 < 30% predicted;
   * Severely reduced diffusion capacity;
   * Baseline hypoxemia and/or hypercapnia;
   * Exercise oxygen consumption < 50% predicted;
   * Severe pulmonary hypertension;
   * Diabetes mellitus with severe end organ damage;
   * Severe cerebral, cardiac, or peripheral vascular disease;
   * Severe chronic heart disease. If the patient has resectable disease but declines surgery after consulting with a thoracic surgeon, he/she will be considered eligible.
6. The patient must have measurable disease.
7. Zubrod Performance Status 0-2;
8. Age ≥ 18;
9. Negative serum or urine pregnancy test within 72 hours prior to registration for women of childbearing potential;
10. Women of childbearing potential and male participants must agree to use a medically effective means of birth control, such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills, throughout their participation in the treatment phase of the study
11. The patient must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Patients with T2 primary tumors > 5 cm or involving the central plural and/or structures of the mediastinum;
2. The primary tumor of any T-stage within or touching the zone of the proximal bronchial tree, defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi);
3. Direct evidence of regional or distant metastases after appropriate staging studies, or synchronous primary malignancy or prior malignancy in the past 2 years except for invasive malignancy that has been treated definitively and the patient remains disease free for > 3 years with life expectancy of > 3 years or carcinoma in situ or early stage skin cancers that have been treated definitively;
4. Previous radiotherapy to the lung or mediastinum;
5. Previous chemotherapy for this lung or mediastinum tumor; chemotherapy for another invasive malignancy is permitted if it has been treated definitively and the patient has remained disease free for > 3 years.
6. Previous surgery for this lung or mediastinum tumor;
7. Plans for the patient to receive other concomitant antineoplastic therapy (including standard fractionated radiotherapy, chemotherapy, biological therapy, vaccine therapy, and surgery) while on this protocol except at disease progression;
8. Patients with active systemic, pulmonary, or pericardial infection;
9. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Videtic, MD, Study Chair — The Cleveland Clinic
Locations (38):
- United States (35):
  - Auburn Radiation Oncology, Auburn, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
- Canada (3):
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Videtic GM, Hu C, Singh AK, Chang JY, Parker W, Olivier KR, Schild SE, Komaki R, Urbanic JJ, Timmerman RD, Choy H. A Randomized Phase 2 Study Comparing 2 Stereotactic Body Radiation Therapy Schedules for Medically Inoperable Patients With Stage I Peripheral Non-Small Cell Lung Cancer: NRG Oncology RTOG 0915 (NCCTG N0927). Int J Radiat Oncol Biol Phys. 2015 Nov 15;93(4):757-64. doi: 10.1016/j.ijrobp.2015.07.2260. Epub 2015 Jul 17. PMID 26530743

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Started | 47 | 47
Eligible | 39 | 45
Started Protocol Treatment (Eligible participants who started protocol treatment) | 39 | 45
Primary Endpoint Population (First 38 eligible participants on each arm who started treatment) | 38 | 38
Peak SUV at 8 Weeks (Eligible participants with peak standardized uptake value (SUV) at baseline and 8 weeks) | 3 | 11
Peak SUV at 1 Year (Eligible participants with peak standardized uptake value (SUV) at baseline and one year) | 4 | 7
Normalized SUV at 8 Weeks (Eligible participants with normalized standardized uptake value (SUV) at baseline and 8 weeks) | 3 | 9
Normalized SUV at 1 Year (Eligible participants with normalized standardized uptake value (SUV) at baseline and one year) | 4 | 7
FEV1 by Best Response (Eligible; FEV1 at baseline and 6 months; complete or partial response, or stable disease) | 26 | 33
DLCO by Best Response (Eligible; DLCO at baseline and 6 months; complete or partial response, or stable disease) | 23 | 28
Completed (Subjects contributing data to results are considered to have completed the study.) | 39 | 45
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 5 | 2
Not completed — RT dose constraints not met | 2 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy) | Total
Number analyzed (Participants) | 39 | 45 | 84
Age, Continuous [Median (Full Range); unit: years] | 75 [57 to 89] | 75 [52 to 87] | 75 [52 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: Counts of ≥ Grade 3 Adverse Events (AE) Graded by CTCAE v4 (Common Terminology Criteria for Adverse Events) That Are Definitely, Probably, or Possibly Related to Treatment (DPPRT)
Description: Number of patients with ≥ grade 3 AE occurring within 1 year of treatment (TRT) start and reported as DPPRT among this subset of CTCAE v4: pericardial effusion, pericarditis, restrictive cardiomyopathy, dysphagia, esophagitis, esophageal fistula/obstruction/perforation/stenosis/ulcer/hemorrhage, rib fracture, brachial plexopathy, recurrent laryngeal nerve palsy, myelitis, atelectasis, bronchopulmonary/mediastinal/pleural/tracheal hemorrhage, bronchial/pulmonary/bronchopleural/tracheal fistula, hypoxia, bronchial/tracheal obstruction, pleural effusion, pneumonitis, pulmonary fibrosis, skin ulceration (thorax only), FEV1 (Forced Expiratory Volume) or FVC (forced vital capacity) decline, or grade 5 related to TRT. Each arm is considered independently. For each arm, >=5 of 38 analyzable subjects experiencing a grade ≥ 3 AE during the 1st year following TRT start would determine the respective TRT excessively toxic. For each arm this design provides 88% power with a 0.10 type I error rate.
Time Frame: From start of treatment to 1 year
Population: First 38 eligible patients per arm who started treatment
Measure: Number; unit: participants
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 38 | 38
participants | 3 | 6

2. Secondary Outcome: 1-year Primary Tumor Control Rate
Description: Primary tumor control is defined as the lack of primary tumor failure. Primary tumor failure is defined as the development of in-field or marginal failure. Primary tumor control time is defined as time from randomization to the the date of primary tumor failure, last known follow-up (censored), or death without failure (competing risk). Primary tumor control rates are estimated using the cumulative incidence method.
Time Frame: From start of treatment to 1 year
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 39 | 45
percentage of participants | 97.1 [85.1 to 99.9] | 97.6 [87.1 to 99.9]

3. Secondary Outcome: 1-year Overall Survival Rate
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method.
Time Frame: From start of treatment to 1 year
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 39 | 45
percentage of participants | 85.4 [70.3 to 93.1] | 91.1 [78.0 to 96.6]

4. Secondary Outcome: 1-year Disease-free Survival Rate
Description: Disease-free survival is defined as being alive without experiencing in-field, marginal, involved lobe, regional or metastatic failure, development of a second primary, or death due to any cause. Disease-free survival time is defined as time from randomization to the the date of first failure or last known follow-up (censored). Disease-free survival rates are estimated using the Kaplan-Meier method.
Time Frame: From start of treatment to 1 year
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 39 | 45
percentage of participants | 78.0 [62.1 to 87.9] | 84.4 [70.1 to 92.3]

5. Secondary Outcome: Change in Peak Standardized Uptake Value (SUV) at 12 Weeks Post-radiotherapy
Description: Standardized uptake value (SUV) describes the level of biologic activity in a particular spot compared to activity elsewhere in the body. An SUV reading of 1 is considered normal cellular activity, with higher values indicating increased activity. Peak SUV is an average SUV computed within a fixed-size volume of interest (VOI), most often containing (and not necessarily centered on) the hottest pixel value. Peak SUV was measured from whole-body FDG-PET (fluorodeoxyglucose - positron emission tomography) scans that were required at baseline and requested (not required) at 12 weeks and 12 months post-radiotherapy. Change from baseline is calculated by subtracting the follow-up value from the baseline value. A positive change from baseline indicates decreased SUV.
Time Frame: Baseline and 12 weeks post-radiotherapy
Population: eligible patients with PET SUV data at at baseline and 12 weeks
Measure: Median (Full Range); unit: SUV
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 3 | 11
SUV | 2.8 [-1.3 to 5] | 1.4 [-3.4 to 10.5]

6. Secondary Outcome: Change in Peak Standardized Uptake Value (SUV) at One Year Post-radiotherapy
Description: Standardized uptake value (SUV) describes the level of biologic activity in a particular spot compared to activity elsewhere in the body. An SUV reading of 1 is considered normal cellular activity, with higher values indicating increased activity. Peak SUV is an average SUV computed within a fixed-size volume of interest (VOI), most often containing (and not necessarily centered on) the hottest pixel value. Peak SUV was measured from whole-body FDG-PET scans that were required at baseline and requested (not required) at 12 weeks and 12 months post-radiotherapy. Change from baseline is calculated by subtracting the follow-up value from the baseline value. A positive change from baseline indicates decreased SUV. SUV does not have a unit.
Time Frame: Baseline and one year
Population: eligible patients with PET SUV data at at baseline and one year
Measure: Median (Full Range); unit: SUV
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 4 | 7
SUV | -0.8 [-5.2 to 2.4] | 3.6 [-1.2 to 12.9]

7. Secondary Outcome: Change in Normalized Standardized Uptake Value (SUV) at 12 Weeks
Description: Standardized uptake value (SUV) describes the level of biologic activity in a particular spot compared to activity elsewhere in the body. An SUV reading of 1 is considered normal cellular activity, with higher values indicating increased activity. SUV was measured from whole-body FDG-PET scans that were required at baseline and requested (not required) at 12 weeks and 12 months post-radiotherapy. Normalized SUV = peak SUV of regions of interest / mean SUV of the aortic arch. Change from baseline is calculated by subtracting the follow-up value from the baseline value. A positive change from baseline indicates decreased SUV. SUV does not have a unit.
Time Frame: Baseline and 12 weeks
Population: eligible patients with normalized SUV at baseline and 12 weeks
Measure: Median (Full Range); unit: SUV
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 3 | 9
SUV | 3.9 [1.1 to 4.2] | 1.4 [-2.5 to 7.2]

8. Secondary Outcome: Change in Normalized Standardized Uptake Value (SUV) at One Year
Description: as for outcome 7
Time Frame: Baseline and one year
Population: eligible patients with normalized SUV at baseline and one year
Measure: Median (Full Range); unit: SUV
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 4 | 7
SUV | 1.0 [-0.7 to 4.1] | 3.9 [-1.6 to 9.4]

9. Secondary Outcome: Change in Percentage of Expected Forced Expiratory Volume in 1 Second (FEV1) by Best Observed Tumor Response at 6 Months Post-radiotherapy [Forced Expiratory Volume in 1 Second (FEV1)]
Description: Forced expiratory volume (FEV1), a measure of pulmonary function, was reported as percentage of the value that would be expected for the normal general population of the same height, age, and sex. Change from baseline is calculated by subtracting the follow-up value from the baseline value. A positive change from baseline indicates decreased FEV1. Best observed tumor response was evaluated using the Revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1 (http://ctep.cancer.gov/protocolDevelopment/docs/recist_guideline.pdf).
Time Frame: From start of treatment to 6 months post-radiotherapy
Population: Eligible patients with FEV1 at baseline and 6 months, and with best tumor response of complete response, partial response, or stable disease
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 26 | 33
percentage of predicted value
  Complete Response: number analyzed (Participants) | 10 | 14
  Complete Response | -2.0 (10.8) | -12.4 (28.0)
  Partial Response: number analyzed (Participants) | 10 | 11
  Partial Response | -0.7 (7.9) | 5.9 (9.0)
  Stable Disease: number analyzed (Participants) | 6 | 8
  Stable Disease | -0.5 (7.6) | -6.1 (11.0)

10. Secondary Outcome: Change in Percentage of Expected Carbon Monoxide Diffusing Capacity (DLCO) by Best Observed Tumor Response at 6 Months Post-radiotherapy
Description: Carbon monoxide diffusing capacity (DLCO), a measure of pulmonary function, was reported as percentage of the value that would be expected for the normal general population of the same height, age, and sex. Change from baseline is calculated by subtracting the follow-up value from the baseline value. A positive change from baseline indicates decreased DLCO. Best observed tumor response was evaluated using the Revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1 (http://ctep.cancer.gov/protocolDevelopment/docs/recist_guideline.pdf).
Time Frame: From start of treatment to 6 months post-radiotherapy
Population: Eligible patients with DLCO at baseline and 6 months, and with best tumor response of complete response, partial response, or stable disease
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 23 | 28
percentage of predicted value
  Complete Response: number analyzed (Participants) | 8 | 12
  Complete Response | 0.1 (23.1) | -2.7 (20.5)
  Partial Response: number analyzed (Participants) | 10 | 11
  Partial Response | 4.1 (9.8) | 2.6 (9.1)
  Stable Disease: number analyzed (Participants) | 5 | 5
  Stable Disease | 12.7 (10.7) | -28.0 (30.6)

11. Secondary Outcome: Association Between Biomarkers and Primary Tumor Control Rate
Time Frame: From start of treatment to 1 year
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Association Between Biomarkers and Grade 2+ Radiation Pneumonitis
Time Frame: From start of treatment to 1 year
Population: as for outcome 11
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Eligible participants who started protocol treatment. Participants experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Single-fraction SBRT (34 Gy) | Multiple-fraction SBRT (48 Gy)
Serious Adverse Events (participants affected / at risk) | 3/39 | 3/45
Other Adverse Events (participants affected / at risk) | 27/39 | 30/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-fraction SBRT (34 Gy) (N=39) | Multiple-fraction SBRT (48 Gy) (N=45)
Heart failure (Cardiac disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-fraction SBRT (34 Gy) (N=39) | Multiple-fraction SBRT (48 Gy) (N=45)
Pericardial effusion (Cardiac disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 7 | 10
Lung infection (Infections and infestations) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 7 | 2
Carbon monoxide diffusing capacity decreased (Investigations) | 5 | 1
Forced expiratory volume decreased (Investigations) | 3 | 2
Vital capacity abnormal (Investigations) | 2 | 1
Weight loss (Investigations) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.